CLINICAL TRIAL: NCT06508671
Title: Effects of DL-3-n-butylphthalide on Chemotherapy-Induced Cognitive Impairment (NBP CICI)：a Prospective, Randomized, Double Blinded, Multicenter, Placebo Controlled Study
Brief Title: Effects of DL-3-n-butylphthalide on Chemotherapy-Induced Cognitive Impairment
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chuansheng Zhao, Professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NBP-CICI-202405
Record Dates: First submitted 2024-07-14; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Chemotherapy-Related Cognitive Impairment; DL-3-n-butylphthalide
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment | interventions — 3-n-butylphthalide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dl-3-n-butylphthalide (Experimental): Take 200 mg butylphthalide soft capsules (NBP) orally three times a day for 24 weeks
  Interventions: Drug: DL-3-n-butylphthalide
- placebo (Placebo Comparator): Take 200 mg placebo of the same appearance with NBP orally three times a day for 24 weeks
  Interventions: Drug: Empty Medication Capsules

INTERVENTIONS:
Drug: DL-3-n-butylphthalide — Take butylphthalide soft capsules orally
  Arms: dl-3-n-butylphthalide
Drug: Empty Medication Capsules — Take empty medication capsules orally
  Arms: placebo

SUMMARY:
Chemotherapy-related cognitive Impairment (CICI) is a series of neurocognitive deficits experienced during and after cancer chemotherapy. Studies have reported that CICI affects 25% to 75% of survivors and can persist for years after chemotherapy is discontinued, causing more severe progressive manifestations and placing a heavy burden on families and society. Numerous studies have proposed several potential mechanisms and etiologies for CICI, including direct neurotoxicity, disruption of the blood-brain barrier, reduced hippocampal neurogenesis, white matter abnormalities, secondary neuroinflammatory responses, and increased oxidative stress. At present, there is no clear and effective diagnosis and therapy for CICI, and how to diagnose and treat cognitive impairment caused by chemotherapy effectively is still the focus and difficulty.

Based on the previous consensus on the application of dl-3-n-butylphthalide, butylphthalein can play a neuroprotective role by reducing oxidative stress and inflammatory response, inhibiting neuronal apoptosis, improving mitochondrial function and other mechanisms, and significantly improve the performance of the central nervous system caused by cerebral ischemia and vascular dementia. However, the increase of neuroinflammatory response and oxidative stress is precisely one of the potential mechanisms of CICI pathogenesis. Therefore, based on the above findings, this study hypothesized that dl-3-n-butylphthalide would also have considerable efficacy in the treatment of CICI.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment with paclitaxel drugs (such as paclitaxel/docetaxel/albumin-based paclitaxel, etc.) or platinum-based chemotherapy (cisplatin), and not combined with other chemotherapy drugs; (Cancer type is not limited)
2. Sign the informed consent and understand the purpose and significance of the study;
3. Aged between 35 and 80 years old;
4. Ability to complete the questionnaire on their own or with assistance;
5. Complaints of cognitive impairment involving memory and/or other cognitive areas lasting for at least 3 months;
6. Cancer treatment has been completed and is considered curable, with the exception of endocrine therapy after chemotherapy;
7. MMSE score: 18-26;
8. Clinical Dementia Rating (CDR) score: 0.5-2;
9. Fluent in Chinese;
10. No visual or hearing impairment;
11. Did not participate in another intervention study within 6 months prior to commencing this study;

Exclusion Criteria:

1. Diagnosed with a cognitively impaired disease, such as Alzheimer's disease;
2. Patients will be excluded from fMRI testing if they are claustrophobic, have MRI contraindications such as pacemakers or metal implants, and patients who did not undergo fMRI testing may still participate in clinical trials if all other enrollment criteria are met;
3. Take medications that may affect cognitive function
4. History of brain metastases or other brain tumors;
5. History of stroke or severe head trauma;
6. History of epilepsy or other seizures;
7. Pregnant or considering becoming pregnant;
8. Any active nervous system or untreated/unremitted mental disorder (such as active major depressive disorder or other major mental disorder described in the DSM-5, allowing treatment of depression if treatment is stable)
9. Any history of alcohol or drug abuse or dependence within the past 2 years;
10. Any major systemic disease or unstable medical condition that may cause difficulty in complying with the protocol, including: a history of myocardial infarction or instability in the past year, serious cardiovascular disease (including angina or congestive heart failure with resting symptoms, or clinically significant abnormalities in the electrocardiogram), clinically significant and/or unstable lung, gastrointestinal, liver or kidney disease;
11. Have taken any non-research drugs to improve cognitive function within 4 weeks prior to enrollment;
12. Have taken butylphthalein in the past 30 days.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mini-mental State Examination (MMSE) | Before chemotherapy,during chemotherapy (12 week after the start of chemotherapy,24 week after the start of chemotherapy),after chemotherapy (12 days after the last chemotherapy)
  The scale ranges from 0 to 30 points. Test scores are closely related to literacy level, and the normal cut-off values are: illiterate >17 points, primary >20 points, junior high school and above >24 points. Combined with the basic characteristics of patients, preoperative and post-chemotherapy assessment was performed to determine the dementia status of patients.
Montreal Cognitive Assessment (MoCA) | Before chemotherapy,during chemotherapy (12 week after the start of chemotherapy,24 week after the start of chemotherapy),after chemotherapy (12 days after the last chemotherapy)
  Patients' cognitive domains were assessed with 11 test items in eight cognitive domains: attention and concentration, executive function, memory, language, visual structure skills, abstract thinking, computation, and orientation. Total score 30, ≥26 normal. Combined with the basic characteristics of patients, preoperative and post-chemotherapy assessment was performed to determine the status of patients with mild cognitive impairment.

SECONDARY OUTCOMES:
Clinician's Interview-based Impression of Change plus caregiver input(CIBIC-plus) | Before chemotherapy,during chemotherapy (12 week after the start of chemotherapy,24 week after the start of chemotherapy),after chemotherapy (12 days after the last chemotherapy)
  CIBIC-plus reflects the clinical improvement of the subject through interviews with the subject and their caregivers.
Clinical Dementia Rating(CDR) | Before chemotherapy,during chemotherapy (12 week after the start of chemotherapy,24 week after the start of chemotherapy),after chemotherapy (12 days after the last chemotherapy)
  CDR is a multidimensional dementia severity scale, scored on a 0-3 scale, with higher scores indicating poorer functioning.
Activities of Daily Living (ADL) | Before chemotherapy,during chemotherapy (12 week after the start of chemotherapy,24 week after the start of chemotherapy),after chemotherapy (12 days after the last chemotherapy)
  ADL are used to assess a patient's ability to perform daily living.
Hamilton Depression Scale(HAMD) | Before chemotherapy,during chemotherapy (12 week after the start of chemotherapy,24 week after the start of chemotherapy),after chemotherapy (12 days after the last chemotherapy)
  HAMD is used to assess the severity and progression of depressive symptoms.
Hamilton Anxiety Scale(HAMA) | Before chemotherapy,during chemotherapy (12 week after the start of chemotherapy,24 week after the start of chemotherapy),after chemotherapy (12 days after the last chemotherapy)
  HAMA is mainly used to assess the severity of neurosis and other anxiety symptoms in patients.
Self-rating depression scale(SDS) | Before chemotherapy,during chemotherapy (12 week after the start of chemotherapy,24 week after the start of chemotherapy),after chemotherapy (12 days after the last chemotherapy)
  SDS is mainly suitable for adults with depressive symptoms, and can intuitively reflect the subjective feelings of depressed patients.
self-rating anxiety scale(SAS) | Before chemotherapy,during chemotherapy (12 week after the start of chemotherapy,24 week after the start of chemotherapy),after chemotherapy (12 days after the last chemotherapy)
  SAS is mainly suitable for adults with anxiety symptoms and can directly reflect the subjective feelings of patients with anxiety.
Functional Magnetic Resonance Imaging(fMRI) | Before chemotherapy,during chemotherapy (12 week after the start of chemotherapy,24 week after the start of chemotherapy),after chemotherapy (12 days after the last chemotherapy)
  fMRI is a research method that stimulates specific senses to cause neural activity (functional area activation) in the corresponding parts of the cerebral cortex and shows it through magnetic resonance images.
Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Before chemotherapy,during chemotherapy (12 week after the start of chemotherapy,24 week after the start of chemotherapy),after chemotherapy (12 days after the last chemotherapy)
  PRO-CTCAE is a tool used to document self-reported adverse events and their severity on a 5-point scale. In our trial, we plan to evaluate 12 symptoms selected from the original PRO-CTCAE scale, specifically decreased appetite, nausea, vomiting, heartburn, bloating, constipation, diarrhea, abdominal pain, insomnia, fatigue, headache, and dizziness.